CLINICAL TRIAL: NCT03310086
Title: Evaluation of the Efficiency of Corticision on Accelerating of Leveling and Alignment Lower Crowded Incisors Using Cone Beam Computed Tomography - A Randomized Controlled Trial
Brief Title: Acceleration of Lower Anterior Teeth Leveling and Alignment Using Corticision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-07-2017
Record Dates: First submitted 2017-10-09; First posted 2017-10-16 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Crowding, Tooth
Keywords: corticision; CBCT; Crowding
MeSH Terms: conditions — Malocclusion; Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional fixed appliance (Experimental): Fixed orthodontic appliances will be applied for aligning and leveling of lower anterior teeth up to 19*25 stainless steel wires using traditional brackets; American Orthodontics Master® MBT 0.022" Brackets
  Interventions: Device: Traditional fixed appliance
- Fixed appliance and corticision (Experimental): Fixed orthodontic appliances with corticison will be applied for aligning and leveling of lower anterior teeth up to 19*25 stainless steel wires using traditional brackets; American Orthodontics Master® MBT 0.022" Brackets
  Interventions: Device: Traditional fixed appliance; Procedure: Corticision

INTERVENTIONS:
Device: Traditional fixed appliance — aligning and leveling of lower anterior teeth using traditional fixed appliance.
Procedure: Corticision — Corticison, cortical bone incision without flap elevation, will be applied to the lower anterior teeth
  Arms: Fixed appliance and corticision

SUMMARY:
This experimental study will evaluate the effect of corticision on accelerating the leveling and alignment of lower crowded incisors compared with the control untreated group using cone beam computed tomography.

The study sample will consist of 26 patients with less than 6 mm crowding. The sample will be allocated randomly into two experimental groups.

The brackets and passive SS wire will be applied with radiographic metal guides between each tooth to allow for accurate corticision site 2 mm below the gingival papilla and to prevent tooth roots injury. The dentoalveolar changes occurring after leveling and alignment of lower anterior teeth will be evaluated using CBCT radiographs, Frequency, degree of root resorption, and the incidence of bone dehiscence will be assessed in relation to initial situation.

DETAILED DESCRIPTION:
Crowding is the most common form of malocclusion. Different methods have been used to resolve crowding, including extraction and nonextraction. Corticision is an important methods to accelerate tooth movement in crowded cases. Cortical bone incision without flap elevation enhances turnover rate of surrounding structures and decreases the time for leveling and alignment. In orthodontics, CBCT imaging has been applied to evaluate impacted teeth and root resorption. But the data are very rare regarding the application of CBCT in tooth movement. So CBCT will be used in this research to evaluate the amount of external apical root resorption (EARR) and presence of dehiscence in the lower anterior teeth in the crowded cases. Furthermore, the duration of alignment will be compared between corticision group and non-corticision group.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18 years or more
* complete permanent dentition with second molars
* crowding of less than 6 mm
* good healthy patients without systematic diseases
* absence of spaces in the lower dental arch
* orthodontic treatment protocol does not required extraoral appliances, intraoral elastics, and expansion during leveling and alignment in the lower arch
* good oral hygiene
* absence of periodontal lesion

Exclusion Criteria:

* patients with syndromes, clefts, or craniofacial abnormalities or systematic diseases
* poor oral hygiene or periodontal lesion
* previous orthodontic treatment.
* Inability for brackets bonding in lower anterior teeth
* presence of extreme skeletal discrepancy in vertical , transverse and anteroposterior relations
* Delay rebonding of any loosing brackets for more than one week in the lower anterior teeth

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Speed of lower teeth movement. | After the leveling and alignment stage of the lower teeth, which will take approximately 9 months
  The speed of lower teeth movement during leveling and alignment stage will be measured and compared between groups.

SECONDARY OUTCOMES:
Changes of lower teeth torque | Changes will be evaluated before and after the lower teeth leveling and alignment stage, which will take approximately 8 months
  The torque changes of the lower teeth will be evaluated and compared between the 2 groups using CBCT.
Changes of lower teeth tipping | Changes will be evaluated before and after the lower teeth leveling and alignment stage, which will take approximately 8 months
  The tipping changes of the lower teeth will be evaluated and compared between the 2 groups using CBCT.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S Burhan, PhD., Study Chair — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Result] Guo QY, Zhang SJ, Liu H, Wang CL, Wei FL, Lv T, Wang NN, Liu DX. Three-dimensional evaluation of upper anterior alveolar bone dehiscence after incisor retraction and intrusion in adult patients with bimaxillary protrusion malocclusion. J Zhejiang Univ Sci B. 2011 Dec;12(12):990-7. doi: 10.1631/jzus.B1100013. PMID 22135148
- [Result] Park YG. Corticision: A Flapless Procedure to Accelerate Tooth Movement. Front Oral Biol. 2016;18:109-17. doi: 10.1159/000351904. Epub 2015 Nov 24. PMID 26599124
- [Result] Ponder SN, Benavides E, Kapila S, Hatch NE. Quantification of external root resorption by low- vs high-resolution cone-beam computed tomography and periapical radiography: A volumetric and linear analysis. Am J Orthod Dentofacial Orthop. 2013 Jan;143(1):77-91. doi: 10.1016/j.ajodo.2012.08.023. PMID 23273363
- [Result] Alikhani M, Raptis M, Zoldan B, Sangsuwon C, Lee YB, Alyami B, Corpodian C, Barrera LM, Alansari S, Khoo E, Teixeira C. Effect of micro-osteoperforations on the rate of tooth movement. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):639-48. doi: 10.1016/j.ajodo.2013.06.017. PMID 24182579
- [Result] Castro IO, Alencar AH, Valladares-Neto J, Estrela C. Apical root resorption due to orthodontic treatment detected by cone beam computed tomography. Angle Orthod. 2013 Mar;83(2):196-203. doi: 10.2319/032112-240.1. Epub 2012 Jul 19. PMID 22812378
- [Result] Mathews DP, Kokich VG. Accelerating tooth movement: the case against corticotomy-induced orthodontics. Am J Orthod Dentofacial Orthop. 2013 Jul;144(1):5-13. doi: 10.1016/j.ajodo.2013.04.008. No abstract available. PMID 23810039